CLINICAL TRIAL: NCT03613246
Title: Clinical Outcomes of the NVT ALLEGRA TAVI System TF in Failing Calcified Aortic Heart Valves in a Real-world Patient Population With Elevated Surgical Risk
Brief Title: NVT ALLEGRA TAVI System TF in Failing Calcified Aortic Heart Valves in a Real-world Patient Population
Acronym: FOLLOW
Status: Active, not recruiting | Type: Observational
Sponsor: NVT GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: NVT04FOL
Record Dates: First submitted 2018-07-06; First posted 2018-08-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Transcatheter Aortic Valve Implantation
Keywords: TAVI; Aortic valve stenosis; ALLEGRA
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients who undergo TAVI for symptomatic severe stenosed aortic heart valves
- Cohort 2:: patients undergoing a VIV procedure in failing surgical bioprostheses.

SUMMARY:
The study collects real-world data of patients who were treated with the ALLEGRA TAVI System TF and evaluates early and midterm clinical and quality of life outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic degeneration of severe calcified aortic heart valve OR failing surgical aortic bioprosthetic valve
2. Acceptable candidate for elective treatment with the ALLEGRA TAVI System TF (according to the most recent version of the ALLEGRA Instructions For Use)
3. High risk for surgery as assessed by the heart team
4. Has signed the Patient Informed Consent Form >= 18 years

Exclusion Criteria:

General:

1. Echocardiographic evidence of intracardiac thrombus or vegetation
2. Significant aortic disease such as severe obstructive calcification or marked tortuosity or kinking which will preclude a safe advancement of the ALLEGRA TAVI System TF
3. Iliofemoral vessel conditions such as severe obstructive calcification, severe tortuosity or kinking that would preclude safe placement of an 18 Fr introducer sheath or make endovascular access to the aortic valve impossible
4. Severe ventricular dysfunction with LVEF <20%
5. Evidence of active endocarditis or other acute infections
6. Renal failure requiring continuous renal replacement therapy
7. Known hypersensitivity to contrast media, which cannot be adequately pre-medicated or contraindication to anticoagulant or anti-platelet medication or to nitinol alloy or to bovine tissue
8. Life expectancy ≤ 12 months due to other medical illness
9. Currently participating in another investigational drug or device study

Patients with native aortic valve disease:

1. Unicuspid or bicuspid aortic valve
2. Non-calcified aortic stenosis
3. Combined aortic valve disease with predominant aortic regurgitation > 3
4. Distance between aortic valve basal plane and the orifice of the lowest coronary artery < 8 mm

Patients with degenerated surgical bioprosthetic aortic valves:

1. Low position of the coronary ostia, especially in combination with shallow sinuses
2. Internal diameter of the bioprosthesis is ≤16 mm or >28 mm
3. Partially detached leaflets that in the aortic position may obstruct a coronary ostium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic patients with elevated surgical risk and candidate for TAVI with severe calcified and stenotic aortic valves or failing surgical bioprosthetic aortic valves.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2029-01-26 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death | 30 days post-index procedure

SECONDARY OUTCOMES:
All-cause mortality | up to five years
Technical success of implantation | day of procedure
  Technical success of implantation, as defined by:
  * absence of procedural mortality AND
  * correct positioning of a single prosthetic heart valve into the proper anatomical location AND
  * no prosthesis - patient mismatch AND
  * mean aortic valve gradient <20 mmHg, AND
  * no moderate or severe prosthetic valve regurgitation
Assesment of NYHA classification | 30 days, 12 month, 24 month, 36 month, 48 month, 60 month
Safety profile according to VARC II | 30 days
  Early Safety
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury-Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure
  Time-related valve safety
  * Structural valve deterioration as defined by
    * Requiring repeat procedure (transcatheter or surgical heart valve replacement)
    * Valve-related dysfunction defined by
      * mean aortic valve gradient ≥20 mmHg and
      * no moderate or severe prosthetic valve regurgitation
  * Prosthetic valve endocarditis
  * Prosthetic valve thrombosis
  * Thrombo-embolic events (e.g. stroke)
  * VARC bleeding, unless clearly unrelated to valve therapy
In-hospital mortality | date of procedure till date of estimated discharge, assessed up to two weeks
Quality of life (EQ5D 5L) | 30 days, 12 month, 24 month, 36 month, 48 month, 60 month
New pacemaker implantation | up to five years
assessment of mean aortic gradient post-implantation | up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schäfer, MD, Principal Investigator — Herz-und Gefäßzentrum Bad Bevensen, Germany
Locations (14):
- Oulu University Hospital, Oulu, Finland
- Germany (5):
  - Herz- und Gefäßzentrum Bad Bevensen, Bad Bevensen
  - Schuechtermann-klinik, Bad Rothenfelde
  - Kath. Marienkrankenhaus, Hamburg
  - MH Hannover, Hanover
  - SLK-Kliniken Heilbronn, Heilbronn
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Clinica Mediterranea Neapel, Naples
- Heartcentre Catharina Hospital Eindhoven, Eindhoven, Netherlands
- Spain (4):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Alvaro Cunqueiro, Vigo
- Morriston Hospital, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No